CLINICAL TRIAL: NCT01073072
Title: Multicentric Prospective Randomized Study Comparing Technique of Tension-free Repair With Placement of a Bovine Pericardium Bioprosthesis (Tutopatch® and Tutomesh®) to Current Conventional Surgical Techniques in Potentially Contaminated Hernia Repair and Abdominal Wall Reconstruction
Brief Title: Study Comparing Tutomesh® Repair to Conventional Surgical Techniques in Potentially Contaminated Hernia Repair and Abdominal Wall Reconstruction
Acronym: Tutomesh
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Régional Universitaire Montpellier (Other)
Responsible Party: Principal Investigator, David Nocca, Dr. David NOCCA, CHRU Montpellier, Centre Hospitalier Régional Universitaire Montpellier
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-A00875-50
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Potentially Contaminated Hernia Repair; Potentially Contaminated Abdominal Wall Reconstruction
Keywords: bovine pericardium bioprosthesis; contamination; hernia repair; abdominal wall reconstruction; Tutomesh; Tutopatch; Potentially Contaminated Hernia Repair; Potentially Contaminated Abdominal Wall Reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tutomesh (Experimental): Technique of abdominal wall reconstruction strengthened by Tutomesh®
  Interventions: Procedure: Technique Tutomesh®
- conventional repair (Active Comparator): Conventional technique to repair incisional or abdominal wall hernias
  Interventions: Procedure: Conventional technique

INTERVENTIONS:
Procedure: Conventional technique — Conventional technique to repair potentially contaminated incisional or abdominal wall hernias
  Arms: conventional repair
Procedure: Technique Tutomesh® — Technique of abdominal wall reconstruction or hernia repair strengthened by Tutomesh® in potentially contaminated environment.
  Arms: Tutomesh

SUMMARY:
This is a multicentric prospective randomized study comparing technique of tension-free repair with placement of a bovine pericardium bioprosthesis (Tutopatch® and Tutomesh®) to current conventional surgical techniques in potentially contaminated hernia repair and abdominal wall reconstruction.

The hypothesis is that using Tutomesh® prostheses reduces the risk of postoperative complications at 30 days in the treatment of incisional hernias or complicated abdominal wall hernias (ref early complications) for potentially contaminated fields.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with an incisional hernia or complicated hernia contraindicating the use of non absorbable mesh:

  * Infected incisional hernia: abdominal wall abscess, chronic fistula
  * Incisional hernia with high septic potential: incisional hernia with strangulation of one or more intestinal loops, repair of incisional hernia during surgery requiring opening of the digestive tube (digestive resection, restoration of digestive continuity, gastro-intestinal perforation, peritonitis from digestive origin)
  * Recurrent incisional hernia with problem of cutaneous healing
  * Incisional hernia requiring important intestinal adhesiolysis
* Patients signing informed consent form after reading and understanding the information letter _ Patients are more than 18 year old

Exclusion Criteria:

* Patient with major anesthetic risk (ASA 4)
* Patient suffering from immunodepression or under immunosuppressor treatment (corticoids…)
* Patients already enrolled in another study
* Patient suffering from severe disease not allowing a 1-year follow-up
* Patient refusing to be enrolled after consulting the information letter
* Patient presenting with a too large incisional hernia, superior to 140x200 mm
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2009-01; Primary Completion 2010-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
risk of postoperative complications: occurrence of complications related to pathology or surgery will be evaluated with the report of adverse events and emergency visits | 30 days

SECONDARY OUTCOMES:
recurrence risk: Assessment of relapse thanks to emergency visits and to adverse events' report | 1 year
the impact on postoperative pain: Assessment of postoperative pain by postponing analgesics | 1 year
the socio-economic impact will be evaluated with the concomitant treatment and hospitalisations. | 1 year
the impact on patients' quality of life: The evaluation of patient's quality of life will be done with the questionnaire quality of life SF12 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David Nocca, Dr, Principal Investigator — University Hospital, Montpellier
Locations (19):
- France (19):
  - CH Aix en Provence, Aix-en-Provence
  - CHU Amiens, Amiens
  - Ch Antibes-Juan les pins, Antibes
  - Clinique de la Casamance, Aubagne
  - CH Avignon, Avignon
  - CHG Beziers, Béziers
  - CHU Jean Verdier, Bondy
  - CHU Fréjus, Fréjus
  - CHU Grenoble, Grenoble - La Tronche
  - Hôpital Nord, Marseille
  - CH St Eloi, Montpellier
  - CHU Nantes, Nantes
  - CHU Archet II, Nice
  - CH Nimes, Nîmes
  - CHU Hôtel Dieu, Paris
  - CH Salon de Provence, Salon-de-Provence
  - CH Hautepierre, Strasbourg
  - CHU Rangueil, Toulouse
  - CHU Trousseau, Tours